CLINICAL TRIAL: NCT01190787
Title: A Multicenter Phase II Study of Subcutaneous Velcade Plus Oral Melphalan and Prdnisone or Plus Cycloposphamide and Prednisone or Plus Prednisone in Newly Diagnosed Elderly Multiple Myeloma Patients
Brief Title: Subcutaneous Velcade Plus Oral Melphalan and Prednisone or Plus Cycloposphamide and Prednisone or Plus Prednisone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Myeloma Network B.V. (Network)
Collaborators: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26866138MMY2069
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Elderly Patients; Diagnosis; Velcade subcutaneous; Prednisone; Melphalan; Cyclophosphamide
MeSH Terms: conditions — Multiple Myeloma; Disease | interventions — Bortezomib; Melphalan; deltacortene; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- VMP (Experimental): INDUCTION Velcade will be given as subcutaneous (SC) injection. Each cycle will be repeated every 28 days.
  Melphalan will be given orally. Each cycle will be repeated every 28 days. Prednisone will be given orally.Each cycle will be repeated every 28 days. MAINTENANCE Velcade will be given a SC injection. Each cycle will be repeated every 28 days.
  Interventions: Drug: velcade subcutaneous melphalan prednisone
- VCP (Experimental): INDUCTION Velcade will be given as subcutaneous (SC) injection. Each cycle will be repeated every 28 days.
  Cyclophosphamide will be given orally. Each cycle will be repeated every 28 days.
  Prednisone will be given orally.Each cycle will be repeated every 28 days. MAINTENANCE Velcade will be given a SC injection. Each cycle will be repeated every 28 days.
  Interventions: Drug: velcade cyclophosphamide prednisone
- VP (Experimental): INDUCTION Velcade will be given as subcutaneous (SC) injection. Each cycle will be repeated every 28 days.
  Prednisone will be given orally.Each cycle will be repeated every 28 days. MAINTENANCE Velcade will be given a SC injection. Each cycle will be repeated every 28 days.
  Interventions: Drug: velcade prednisone

INTERVENTIONS:
Drug: velcade subcutaneous melphalan prednisone — INDUCTION Velcade will be given as subcutaneous (SC) injection. Each cycle will be repeated every 28 days.
  Melphalan will be given orally. Each cycle will be repeated every 28 days. Prednisone will be given orally.Each cycle will be repeated every 28 days. MAINTENANCE Velcade will be given a SC injection. Each cycle will be repeated every 28 days.
  Other Names: Bortezomib, Alkeran, Deltacortene
  Arms: VMP
Drug: velcade cyclophosphamide prednisone — INDUCTION Velcade will be given as subcutaneous (SC) injection. Each cycle will be repeated every 28 days.
  Cyclophosphamide will be given orally. Each cycle will be repeated every 28 days.
  Prednisone will be given orally.Each cycle will be repeated every 28 days. MAINTENANCE Velcade will be given a SC injection. Each cycle will be repeated every 28 days.
  Other Names: Bortezomib,Endoxan, deltacortene
  Arms: VCP
Drug: velcade prednisone — INDUCTION Velcade will be given as subcutaneous (SC) injection. Each cycle will be repeated every 28 days.
  Prednisone will be given orally.Each cycle will be repeated every 28 days. MAINTENANCE Velcade will be given a SC injection. Each cycle will be repeated every 28 days.
  Other Names: Bortezomib, deltacortene
  Arms: VP

SUMMARY:
This protocol is a single-arm, three-cohort, phase II multicenter study designed to assess the safety and the efficacy of three all-oral combinations: Velcade with continuous low-dose melphalan and prednisone (VMP) or with continuous low-dose cyclophosphamide and prednisone (VCP) or Velcade with low-dose prednisone could be effective and well tolerated (VP).

DETAILED DESCRIPTION:
This protocol is a single-arm, three-cohort, phase II multicenter study designed to assess the safety and the efficacy of VMP and VCP and VP as up-front treatment in elderly MM patients. The combination of weekly subcutaneous administrations of Velcade with continuous low-dose melphalan and prednisone (VMP) or with continuous low-dose cyclophosphamide and prednisone (VCP) or Velcade with low-dose prednisone could be effective and well tolerated (VP).

Patients will be evaluated at scheduled visits in up to 3 study periods: pre-treatment, treatment and long-term follow-up (LTFU).

The pre-treatment period includes screening visits, performed at study entry. After providing written informed consent to participate in the study, patients will be evaluated for study eligibility. The screening period includes the availability of inclusion criteria described above.

The treatment period includes induction and maintenance.

Subjects receive:

1. Induction therapy:

   nine 4-week courses of Velcade/Melphalan/Prednisone (VMP) or nine 4-week courses of Velcade/Cyclophosphamide/Prednisone (VCP) or Nine 4-week courses of Velcade/Prednisone (VP).
2. Maintenance therapy:

Velcade alone During the induction period patients will attend periodic study centre visits each scheduled Velcade administration in order to asses the toxicity and efficacy of the treatment. During the maintenance period, all patients will attend study centre visits every 4 weeks, until development of confirmed PD. The response will be assessed after each cycle.

During the LTFU period, after development of confirmed PD, all patients are to be followed for survival during the LTFU period every 3 months via telephone or office visit.

The duration of treatment period, including the maintenance treatment is approximately 3 years. The duration of LTFU is approximately 2 years, for a total of 5 years. the occurance of PD will determine the duration of progression-free survival of each patient(secondary objective). The occurrence of death will determine the duration of overall survival (secondary objective).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years old or age < 75 years with abnormal cardiac, pulmonary, renal or hepatic function (unsuitable for protocol with standard inclusion/exclusion criteria).
* Patient is, in the investigator(s) opinion willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Male patient agrees to use an acceptable method for contraception (i.e., condom or abstinence) during study drug therapy (including dose interruption) and for 4 weeks after discontinuation of Velcade therapy.
* Female patient is either post-menopausal for 24 consecutive months or surgically sterilised or agree to continuous abstinence from heterosexual sexual contact or willing to use two acceptable method of birth control at the same time (one highly effective method and one additional effective method) (Highly Effective Methods: Intrauterine device -IUD-; Hormonal -birth control pills, injections, implants-; tubal ligation; partner's vasectomy; Additional Effective Methods: Latex condom; Diaphragm; Cervical Cap) for 4 weeks prior to beginning study drug therapy, during study drug therapy (including dose interruption) and for 4 weeks after discontinuation of therapy.
* Patient was a newly diagnosed multiple myeloma based on standard criteria
* Patient has measurable disease, defined as follows:
* Secretory myeloma: any quantifiable serum monoclonal protein value (generally, but not necessarily, greater than 1 g/dL of IgG M-Protein and greater than 0.5 g/dL of IgA M-Protein) and, where applicable, urine light-chain excretion of >200 mg/24 hours;
* Non-secretory myeloma: > 30% plasma cells in the bone marrow and at least one plasmacytoma > 2 cm as determined by clinical examination or applicable radiographs (i.e., MRI or CT scan).
* Patient has a Karnofsky performance status > 50%.
* Patient has a life-expectancy >3 months
* Pretreatment clinical laboratory values within 14 days of enrolment:
* platelet count ≥ 80x109/L
* hemoglobin ≥ 8 g/dL
* absolute neutrophil count (ANC) ≥ 1.0x109/L
* AST ≤ 2.5 times the upper limit of normal
* ALT ≤ 2.5 times the upper limit of normal
* total bilirubin ≤ 1.5 times the upper limit of normal
* cleareance creatinine ≥ 20 ml/min

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality or psychiatric illness that prevented the subject from signing the informed consent form or placed the subjects at unacceptable risk.
* Previous treatment with anti-myeloma therapy (does not include radiotherapy, bisphosphonates, or a single short course of steroid; < to the equivalent of dexamethasone 40 mg/day for 4 days).
* Pregnant or lactating females
* Known positive for HIV or active infectious hepatitis type A, B or C
* Peripheral neuropathy or neuropatic pain grade 2 or higher, as defined by National Cancer Institute Common Toxicity Criteria (NCI CTC) 3.0
* Infiltrative pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Very Good Partial Response, Complete response rate , Partial response rate | 5 years

SECONDARY OUTCOMES:
Progression free survival | 5 years
Time to progression | 5 years
Time to Next Therapy | 5 years
Overall survival | 5 years
Time to response | 5 years
Duration of response | 5 years
Response rate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mario Boccadoro, MD, Principal Investigator — Fondazione EMN Italy Onlus
Locations (1):
- A.O.U. Città della Salute e della Scienza di Torino - SC Ematologia U, Torino, Italy

REFERENCES:
- [Derived] Montefusco V, Gay F, Spada S, De Paoli L, Di Raimondo F, Ribolla R, Musolino C, Patriarca F, Musto P, Galieni P, Ballanti S, Nozzoli C, Cascavilla N, Ben-Yehuda D, Nagler A, Hajek R, Offidani M, Liberati AM, Sonneveld P, Cavo M, Corradini P, Boccadoro M. Outcome of paraosseous extra-medullary disease in newly diagnosed multiple myeloma patients treated with new drugs. Haematologica. 2020 Jan;105(1):193-200. doi: 10.3324/haematol.2019.219139. Epub 2019 Jun 20. PMID 31221778
- [Derived] Palumbo A, Bringhen S, Mateos MV, Larocca A, Facon T, Kumar SK, Offidani M, McCarthy P, Evangelista A, Lonial S, Zweegman S, Musto P, Terpos E, Belch A, Hajek R, Ludwig H, Stewart AK, Moreau P, Anderson K, Einsele H, Durie BG, Dimopoulos MA, Landgren O, San Miguel JF, Richardson P, Sonneveld P, Rajkumar SV. Geriatric assessment predicts survival and toxicities in elderly myeloma patients: an International Myeloma Working Group report. Blood. 2015 Mar 26;125(13):2068-74. doi: 10.1182/blood-2014-12-615187. Epub 2015 Jan 27. PMID 25628469